CLINICAL TRIAL: NCT07118124
Title: Pediatric Adhesion and New Dermal Approach Study (PANDA)
Brief Title: Pediatric Adhesion and New Dermal Approach Study
Acronym: PANDA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: iRhythm Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: iRT-001-2025
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Syncope; Pediatric; Congenital Athymia; Congenital Heart Disease; Arrhythmia; Arrhythmia in Children
Keywords: Pediatrics; PANDA Study; Zio monitor; Children; arrhythmia in children
MeSH Terms: conditions — Syncope; Heart Defects, Congenital; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single-arm study to analyzable time for use in pediatric patients up to 14 days (Other): Zio monitor
  Interventions: Device: Zio monitor

INTERVENTIONS:
Device: Zio monitor — Evaluate analyzable time of the Zio monitor over the wear duration of up to 14 days in a pediatric population.

SUMMARY:
The purpose of this study is to see if the Zio® monitor device can be worn by children for up to 14-days and to determine if the skin preparation process will provide good adherence to the skin and clear signal quality. The Zio® monitor (Study Device) is an adhesive patch that is worn on the upper left chest for a specified period of time and is similar to a band aid. The Study Device contains a battery-powered heart monitor and will look at the heart rhythm and rate.

DETAILED DESCRIPTION:
This is a prospective single-arm study to demonstrate adequate analyzable time for use in pediatric patients up to 14 days of device wear. The study will incorporate a simplified skin preparation procedure. The objective is to evaluate analyzable time of the Zio® monitor device over the wear duration (up to 14 days) in a population 1 to 17 years of age. The study will incorporate a simplified skin preparation procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Child is <18 years of age and ≥1 year of age and weighing >10 kg (22 pounds) at the time of device application.
2. Child's legally authorized representative is willing and able to provide informed consent and be able to assist the Child in completing all visits for the study. If the Child is old enough to provide assent, it will also be captured.
3. The prescribed Zio monitor wear time is planned to be up to 14 days.

Exclusion Criteria:

1. Child has a known allergy to adhesives or hydrogels or with family history of adhesive skin allergies.
2. Child has a visible skin injury or broken skin at location for study device placement.
3. Child has skin damage and a discharge of clear fluid or pus at the location for study device placement.
4. Child is unable or unwilling to participate or comply with study protocol.
5. The local Investigator deems the Child has a condition that could limit the Child's ability or willingness to participate in the study, or ability to comply with study required procedures and/or follow-up visits. (It is understood that younger age groups of children may present development behavioral challenges in compliance with use of medical devices. Normal development stage should not be considered a reason for exclusion).
6. The child has experienced symptomatic episodes where instance variations in cardiac performance could result in immediate danger to the child or when real-time or in-patient monitoring should be prescribed.
7. Child has an external or wearable cardiac defibrillator or may be exposed to high frequency surgical equipment near strong magnetic fields or devices such as MRI during the wear period.
8. Child has a neuro-stimulator, as it may disrupt the quality of ECG data.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Performance Objective | Up to 14 days
  The duration of non-artifact ECG signal as a proportion of the device total wear time will be assessed. The sample proportion with analyzable time >80% is assumed to be 90%. The performance objective will be met if the lower bound of the 95% confidence interval is at least 75%. Percent analyzable time is defined as the duration of non-artifact ECG signal as a proportion of the device total wear time.

OTHER OUTCOMES:
Safety Measures | From enrollment to the end of the device wear period
  The proportion of participants that experience clinically significant skin irritation during wear will be assessed via a skin irritation assessment performed by the healthcare provider. All adhesive-based wearable devices may lead to skin irritation. Minor itching and redness are expected. Skin reaction during wear should be reported as an adverse event. Adverse events will be reported and assessed for severity and relationship to the study device.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Berul, MD, Principal Investigator — Children's National Research Institute
Locations (4):
- United States (4):
  - Children's National Hospital, Washington D.C., District of Columbia
  - St. Luke's Children's Hospital, Boise, Idaho
  - Boston Children's Hospital, Boston, Massachusetts
  - WashU Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No